CLINICAL TRIAL: NCT00837278
Title: Maternal Serum Cytokine Levels and Angiogenic Factor Levels in Singleton IVF Pregnancies vs Spontaneously Conceived Pregnancies
Brief Title: Maternal Serum Cytokine Levels and Angiogenic Factor Levels in IVF vs Spontaneously Conceived Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MemorialCare (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Kenneth Chan, MD, MemorialCare
Other Study IDs: IVF cytokines; MHS IRB No. 525-08
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Infertility
Keywords: IVF; angiogenic factors; cytokines
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood draws are to be performed at four times. These are 10-15 weeks, 22-28 weeks, 34-40 weeks, and 4-8 weeks postpartum. Additionally, placental biopsies and umbilical cord blood specimens are to be collected for possible future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 IVF: Pregnancies conceived with the use of assisted reproductive technologies. This is defined as a pregnancy conceived with all gametes being handled outside of the body.
- 2 Control: Spontaneously conceived pregnancies.

SUMMARY:
The objective of the study is to compare maternal levels of cytokines and angiogenic factors in IVF vs spontaneously conceived singleton pregnancies. The null hypothesis is that there will be no significant difference.

DETAILED DESCRIPTION:
IVF subjects: Subjects will be screened for participation at the Magella Office in Long Beach. Healthy patients with singleton pregnancies conceived with ART will be invited to participate.

Control subjects: A group of control subjects with spontaneously conceived, singleton pregnancies matched for age, parity, and race, will be identified at our Magella offices in Long Beach.

Sample size: 20 IVF subjects and 20 control subjects will be enrolled. A power analysis was performed using an alpha error of 0.05 and beta error of 0.80. Calculations were made for a 30% difference in the most studied markers during each trimester. The specific markers used in the power analysis were VEGF, sFlt, sEng, PlGF, IL-6, IL-8, TGF-beta1, and TNF-alpha. Using the values for the markers with the most stringent criteria it was determined that 15 patients would be required in each group to demonstrate a significant difference using a p value of 0.05. In anticipation of a 20-25% drop out rate, 20 subjects will be enrolled in each arm.

Specimens will be obtained at the specified intervals. Venipuncture will be performed and no more than 20 ml of blood will be obtained.

Within 2 hours of the blood draw, the blood will be spun at 2000 rpm for 10 minutes. The plasma layer will then be collected into 1 ml aliquots and stored frozen at -80°C. Upon completion of specimen collection, assays will be performed by personnel who are unaware of the outcome of the pregnancy. The markers being evaluated are not currently routinely used in clinical practice thus preventing a retrospective analysis.

The cytokine analysis and VEGF measurements will be performed using Cytokine 29 Plex Kit Premixed Beads, HCYTO-60K-PMX29 (Linco Research, St. Charles, MO, USA). This kit measures various markers and proteins of the immune system to determine the degree of inflammation. Cytokines measured with the kit include: Human IL-1, Human IL-2, Human IL-1ra, Human IL-4, Human IL-5, Human EGF, Human IL-6, Human IL-7, Human TGF,_Human Fractalkine, Human IL-8, Human IL-10, Human IL-12p70, Human IL-13, Human IL-15, Human IL-17, Human IL-1, Human IFNgamma, Human G-CSF, Human GM-CSF, Human TNF, Human Eotaxin, Human MCP-1, Human sCD40L, Human IL-12p40, Human MIP-1, Human MIP-1beta, Human IP-10, and Human VEGF.

The assays will be run according to the established protocol using the 96 well plate provided. Briefly, each serum sample is to be incubated with cytokine microbeads for 1 hour at room temperature. After washing two times, the beads will be incubated with detection antibodies for 30 min. The beads will then be combined with streptavidin-phycoerythrin and remain at room temperature for an additional 30 minutes. After two additional washings, the beads will be resuspended in assay buffer for five minutes and then the beads are to be read on the Luminex Instrument.

Commercially available enzyme-linked immunosorbent assays (ELISAs) for sFlt 1 (BioSource™) (Invitrogen Corporation, Carlsbad, CA), endoglin (R&D Systems Inc, Minneapolis, MN), PIGF (R&D Systems, Inc. Minneapolis, MN) will be used according to established protocols. Briefly, various samples for ELISA measurement will be diluted in respective calibrator diluent. After adding assay diluent, the diluted sample will be placed in a 96-well plate precoated with captured antibodies directed against human sFlt-1, human endoglin, or PlGF, and the plates were incubated for 2 hours. The wells will be washed 4 times in wash buffer and incubated with secondary polyclonal antibody against sFlt-1, endoglin, and PIGF conjugated to horseradish peroxidase for an additional 2 hours. The plates are then washed 4 times in wash buffer.

Substrate solution containing hydrogen peroxide and tetramethylbenzidine will then be added to each well and incubated for 30 minutes under protection from light with stop solution was added to each well also. The optical density will then be determined by subtracting readings at 540 nm from the reading at 450 nm. Protein levels will be calculated using a standard curve derived from a known concentration of respective recombinant proteins. The minimum detectable doses in the assay for sFlt-1, endoglin, and PlGF are 3.5, 7, and 5 pg/mL, respectively. Intraassay and interassay coefficients of variation of 3.5% and 5.5%, respectively, for sFlt-1, 3.2% and 6.5%, respectively, for endoglin, and 6% and 11%, respectively for PlGF.

Following delivery placental biopsies will be obtained for possible further analysis in anticipation of extramural funding pending the results of this study. For each placenta, three small full-thickness samples approximately 2 cm x 2 cm x 2 cm, not to include fetal membranes, will be obtained and stored in a -80ºC freezer pending mRNA extraction. We will follow a standard protocol for placental tissue harvest. The remainder of the placentas will be disposed of per routine on the Labor and Delivery unit.

Additionally, umbilical artery blood will also be obtained following delivery for possible further analysis. Within 2 hours of the blood collection, the blood will be spun at 3000 rpm for 10 minutes. The plasma layer will then be collected into 1ml aliquots and frozen in a -80ºC freezer.

For each subject, maternal demographic information including age, ethnicity, infertility history, previous obstetrical history, pregnancy complications and delivery outcomes will be collected. In addition, neonatal outcome data will be collected including delivery data, birth weight, and complications. See attached data sheet (Appendix B).

All specimens and data from the medical record will be collected and assigned a unique case number. Identifying information (e.g. name, birth date, and medical record number) will not be present in this database. In order to enable us to retrieve the medical record in the future for data verification, a key relating case numbers and medical record numbers will be kept separately. This key will be password protected, with the password only known to the investigators.

With the above exceptions, throughout the course of their pregnancy study participants will receive standard prenatal care as determined by their physicians.

Data Analysis

Categorical data will be analyzed using the Fisher exact test and chi squared test. Student t test and Mann-Whitney U tests will be used for the evaluation of parametric and non parametric continuous data, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with singleton pregnancies conceived with ART and control subjects with spontaneously conceived pregnancies. Only subjects that are already pregnant and have confirmed singleton intrauterine pregnancies are eligible.

Exclusion Criteria:

* Subjects with hypertension, diabetes, renal disease, illicit drug use, tobacco use, morbid obesity, collagen vascular disease, and autoimmune diseases will be excluded from participation.
* Pregnancies that had more than one gestation viewed on ultrasound at any time will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy patients with singleton pregnancies conceived with ART. Only subjects that are already pregnant and have confirmed singleton intrauterine pregnancies are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-03 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
sFlt, human endoglin, PlGF, VEGF, IL-1, IL-2, IL-1ra, IL-4, IL-5, EGF, IL-6, Human IL-7, TGF, Fractalkine, IL-8, IL-10, IL-12p70, IL-13, IL-15, IL-17, IL-1, IFN-gamma, G-CSF, GM-CSF, TNF, Eotaxin, MCP-1, sCD40L, IL-12p40, MIP-1, MIP-1ß, IP-10 | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chan, MD, Principal Investigator — MemorialCare
Locations (1):
- MemorialCare, Long Beach, California, United States